CLINICAL TRIAL: NCT02245958
Title: A Retrospective Chart Review of BOTOX® and Xeomin® for the Management of Cervical Dystonia and Blepharospasm
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-US-NEU-0271
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Cervical Dystonia; Blepharospasm
MeSH Terms: conditions — Torticollis; Blepharospasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BOTOX®: Retrospective chart review of doses of BOTOX® (onabotulinumtoxinA) used as standard of care in clinical practice. No treatment (intervention) was administered.
  Interventions: Other: No Intervention
- Xeomin®: Retrospective chart review of doses of Xeomin® (incobotulinumtoxinA) used as standard of care in clinical practice. No treatment (intervention) was administered.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No treatment (intervention) was administered.

SUMMARY:
This study is a retrospective chart review to evaluate the doses of botulinum Type A toxins BOTOX® (onabotulinumtoxinA) and Xeomin® (incobotulinumtoxinA) used for the treatment of Cervical Dystonia and Blepharospasm in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary diagnosis of idiopathic cervical dystonia or blepharospasm for at least 2 years
* Treatment with Xeomin® and BOTOX® for at least 2 years each.

Exclusion Criteria:

* Having a neuromuscular junction transmission disorder or taking any medications that could affect neuromuscular junction transmission
* Previous surgical procedure involving bone or muscle for the management of cervical dystonia or blepharospasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with cervical dystonia or blepharospasm previously treated with Xeomin® and BOTOX® in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Dose of Botulinum Toxin Used to Treat Cervical Dystonia | 4 Years
Dose of Botulinum Toxin Used to Treat Blepharospasm | 4 Years

SECONDARY OUTCOMES:
Botulinum Toxin Inter-injection Intervals | 4 Years
Number of Participants with Adverse Events | 4 Years
Annual Botulinum Toxin Dose per Patient | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Colonia Roma Z.P., Mexico
- Wakefield, United Kingdom